CLINICAL TRIAL: NCT04014985
Title: Study of Biological Parameters in 100 Girls With RETT Syndrome
Brief Title: Patients With RETT Syndrome
Acronym: RETT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-30; 2018-A01066-49 (Registry Identifier: ANSM)
Record Dates: First submitted 2019-06-06; First posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Rett Syndrome
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Girls with RETT syndrome (Other): 100 girls over 18 years old with RETT syndrome
  Interventions: Other: An extensive biological assessment

INTERVENTIONS:
Other: An extensive biological assessment — To study the morphology of red blood cells, the markers of oxidative stress and the signaling pathway of IFGF1.

SUMMARY:
It was proposed to the French Association of Rett Syndrome (AFSR) to perform an extensive biological assessment in a series of 100 girls with Rett's syndrome and carriers of a mutation in the MECP2 gene in order to confirm or confirm to reverse the abnormalities identified previously and possibly, to highlight new biomarkers of the pathology. The analysis will focus on classical hematological criteria, iron markers, endocrine assays, lipid quantification and markers of inflammation. At the end of the project, each family will receive the complete biological assessment carried out on their daughter which will represent a direct benefit of the implication in this clinical research project.

DETAILED DESCRIPTION:
The MECP2 (Methyl-CpG binding protein) gene, located on the X X28 chromosome, encodes a heterochromatin nuclear protein. Mecp2 is preferentially found in neurons at a postmitotic stage where it promotes brain development. Its ability to fix methylated DNA and contribute to the formation of a transcriptional repression complex attributes this protein to a crucial role in the control of gene expression. However, until today, its exact role is not known. In humans, mutations in the MECP2 gene are at the origin of neurological diseases, the main one being Rett's syndrome (RTT-MIM # 312750) where a mutation of MECP2 is found in 95% of cases. This dominant pathology linked to the X chromosome has a prevalence of 1/10000 to 1/15000 births and affects mostly girls. The course of the pathology is characterized by a cessation of development between 6 and 18 months after birth. Patients present a set of characteristic signs including regression of acquired abilities, manual stereotyping, loss of language, behavioral disorders and severe intellectual disability. In their attempt to better understand the pathology, many laboratories are currently trying to identify abnormal biological parameters in patients that are easy to identify in a non-invasive or minimally invasive way in order to indirectly evaluate the progression of the pathology and to identify biochemical disorders amenable to direct pharmacological intervention.

In autumn 2015, several factors were identified as deregulated in model mice or RTT patients (Rett syndrome). They could be related to the severity of the disease and indicators of its progression. Among these we can mention:

* major structural damage to red blood cells;
* Inflammation demonstrated and challenged ;
* high oxidative stress markers; lipid deregulation and in particular cholesterol abnormalities;
* a deficiency of the signaling pathway of insulin and IGF-1.

ELIGIBILITY:
Inclusion Criteria:

* People with Rett syndrome related to MECP2 gene mutation
* Aged under 18 years old.
* Regularly followed as part of their illness by Prof. Bahi-Buisson in Necker or Pr Milh in Marseille.
* Whose state of health justifies a blood test (dosage of one or more anti-epileptics, recommended annual phosphocalcic balance, pre-therapeutic assessment before introduction of a new molecule ...)
* Whose at least one parent (or legal representative) has signed the consent
* Patient fasting for 6 hours at the time of sampling.

Exclusion Criteria:

* Contraindication to a balance sheet
* Absence of consent of the legal representatives

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of red blood cell morphology | 1 day
  Identification of abnormal red blood cells
Comparison of oxydative stress markers | 1 day
  Identification of abnormally high cytokine levels
Comparison of cholesterol levels | 1 day
  Identification of hight cholesterol levels

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France